CLINICAL TRIAL: NCT03563196
Title: Comparison Of Lung Ultrasound To Chest Radiography For Diagnosis Of Pulmonary Complications After Cardiac Surgery In Children
Brief Title: Diagnosis Of Pulmonary Complications After Cardiac Surgery In Children
Status: Completed | Type: Observational
Sponsor: Shahid Gangalal National Heart Centre (Other)
Responsible Party: Sponsor
Other Study IDs: SGNHC9
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Children; Cardiac Surgery; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chest Radiograph: All the patients will undergo routine chest radiogram on day 1 after operation
  Interventions: Radiation: Chest Radiograph
- Lung Ultrasound: The same patient will undergo ultrasound evaluation of lungs on day 1 after operation
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Radiation: Chest Radiograph — Chest radiogram will be obtained on day 1
  Groups: Chest Radiograph
Diagnostic Test: Lung Ultrasound — Lung ultrasound will be done on day 1
  Groups: Lung Ultrasound

SUMMARY:
Pulmonary complications are frequent in cardiac surgery, representing an important cause of morbidity, prolongation of hospital stay and need for repeated examinations.Chest X-rays are done routinely and even multiple times to detect such complications.Lung ultrasonography is an alternative test to detect pulmonary complications that can be done easily on bedside. Regularly done Chest X-ray exposes patient to ionizing radiation which can be reduced with ultrasonography. Lung ultrasound is gaining popularity in recent years as a non-invasive,radiation-free tool for the diagnosis of various acute and chronic pulmonary diseases due to its bedside convenience, accuracy, and free of radiation.There is increasing evidence to support the use of Lung ultrasound in acute care setting and post-cardiac surgical patients are also considered critically ill. The purpose of this study is to compare diagnostic performance of lung ultrasound in comparison to chest X-ray to detect pulmonary complication after cardiac surgery in children.

DETAILED DESCRIPTION:
Study type: Comparative Study design: Non-randomized,all patients will undergo both ultrasound and chest Xray.

Model:cohort time perspective: prospective Sampling method: non-probability sample Study population: Children less than 14 years Sample size: 54 Place of Study-Shahid Gangalal national Heart Center, Surgical intensive care unit Duration of study: six months Hypothesis: Chest X-ray and Lung ultrasound are equally effective in detecting postoperative pulmonary complications

Inclusion criteria:

Patients after undergoing cardiac surgery who are age below 14 years on post-operative Day 1.

Exclusion criteria Patient's /Guardians' refusal IMAGING PROTOCOL AND TECHNIQUE Following institutional review board approval, a written informed consent will be obtained from all the patients meeting the inclusion criteria before undergoing surgery on pre-operative visit before enrollment in the study.

Lung Ultrasound will be done on the first post-operative day of cardiac surgery and will be compared to Chest X-ray done on the same day for any pulmonary complications . Lung ultrasound examination will be performed by radiologist to detect pleural effusion, consolidation, pulmonary atelectasis, pneumothorax and pulmonary congestion, using Siemens AUCUSON Freestyle Diagnostic Ultrasound System L13-5 linear probe. The transthoracic Lung ultrasound approach will be done in supine and both lateral decubitus positions of the anterior lung area (between the sternum and the anterior axillary line), lateral lung area (between the anterior and posterior axillary lines), and posterior lung area (between the posterior axillary line and the spine) in caudo-cranial direction. Longitudinal, transverse and oblique scans will be included. A routine plain chest radiograph will be obtained in each patient on the same day before performing ultrasound which will be evaluated by an intensivist to detect pleural effusion, consolidation, pulmonary atelectasis, pneumothorax. Both the radiologist and intensivist will be blinded to each other's findings. Comparison of the findings will be done at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged less than 14 years scheduled for cardiac surgery in Shahid Gangalal National Heart Center

Exclusion Criteria:

* guardian's refusal

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged less than 14 years scheduled for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pulmonary complications; Pleural effusion;lung consolidation,lung collapse,pneumothorax | 24 hours
  The ultrasound image of pleural effusion is measured by depth of echo-free space between the visceral and parietal pleura.
  The pulmonary ultrasonic signs of lung consolidation included a hypo-echoic area of varying shape and size with irregular margins of heterogeneous echogenicity and also included dynamic air bronchograms.
  The main features of atelectasis on LUS included lung consolidation and static air bronchograms.
  The ultrasound findings of pneumothorax included absent lung sliding and B lines and so are the comet tail artifacts from the pleura

CONTACTS AND LOCATIONS:
Overall Officials: smriti M bajracharya, MD, Principal Investigator — Registrar in Cardiac Anesthesia and ICU
Locations (1):
- Shahid Gangalal National Heart Center, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided